CLINICAL TRIAL: NCT06437886
Title: Postoperative Recovery After Cardiac Surgery A Randomised Controlled Trial of High-dose Opioid Versus Opioid-sparing Anaesthesia
Brief Title: High-dose Opioid Versus Opioid-sparing Anaesthesia in Cardiac Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yan Fuxia, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-2323
Record Dates: First submitted 2024-05-22; First posted 2024-05-31 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Surgery Patients

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pecto-intercostal fascial block and rectus sheath block-based opioid-sparing anesthesia (Experimental)
  Interventions: Other: opioid-sparing protocol
- high-dose opiod traditional anesthesia (No Intervention)

INTERVENTIONS:
Other: opioid-sparing protocol — Patients in the OSA group was administrated with 0.5 to 1 mcg·kg-1 sufentanil and received PIFB combined with RSB after anesthetic induction. Patients in the control group were recommended to receive 2 to 3 mcg·kg-1 opioid-based sufentanil. PIFB was conducted at the T2 to T5 levels under ultrasound guidance. Each side received 20 ml 0.3% ropivacaine containing 2.5 mg dexamethasone. Bilateral RSB was conducted after the PIFB and the needle was inserted into the plane between the rectus abdominal muscle and its posterior sheath using an in-plane approach. After verifying needle placement, 15 ml 0.3% ropivacaine containing 2.5 mg dexamethasone was delivered to each side. In the control group, patients received no procedure and were administrated with traditional anesthetic protocol. Patients received continuous intravenous sufentanil (50 to 100 mg) and tropisetron (5 to 10 mg) at 2 ml·h-1 for the first 48 hours after surgery.
  Arms: pecto-intercostal fascial block and rectus sheath block-based opioid-sparing anesthesia

SUMMARY:
BACKGROUND In cardiac surgery, high-dose opioid contributes to adverse events associated with poor postoperative outcomes. There is growing evidence that nerve block-based multi-modal anesthesia protocols may reduce intraoperative opioid consumption without compromising analgesia management and consequently improve patient's early postoperative recovery.

OBJECTIVE To determine whether opioid-sparing anaesthesia based on ultrasound-guided nerve block could improve early postoperative recovery after cardiac surgery.

DESIGN A randomised controlled trial. SETTING A tertiary hospital. PATIENTS Eighty patients aged 45 to 70 years undergoing cardiac surgery were enrolled. Key exclusion criteria included contraindication to interventions or drugs and a history of chronic pain or chronic opioid use.

INTERVENTIONS Eligible patients were randomised at a 1:1 ratio to receive either opioid-sparing anaesthesia based on ultrasound-guided nerve block (intervention group) or opioid-based anaesthesia (control group).

MAIN OUTCOME MEASURES The primary outcome was the global score of the 15-item Quality of Recovery (QoR-15) questionnaire at 24h after surgery. Secondary outcomes included QoR-15 at 72h after surgery, postoperative pain score, the incidence of postoperative adverse events and chronic pain. Other outcomes included endotracheal intubation duration, length of hospitalization, and hospital costs.

ELIGIBILITY:
Inclusion Criteria:

Male or female adult patients aged 45 to 70 years, awaiting elective cardiac surgery, and American Society of Anaesthesiologists physical status classes II or III were eligible.

Exclusion Criteria:

contraindications to punctual or local anesthetic drugs, a history of chronic pain or chronic opioid use, and an inability to communicate or refuse to enroll.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-07-22 (Estimated); Study Completion 2024-07-22 (Estimated)

PRIMARY OUTCOMES:
QoR-15 at 24h | at 24 hours after surgery
  the global score of the 15-item Quality of Recovery (QoR-15) questionnaire at 24h after surgery

SECONDARY OUTCOMES:
QoR-15 at 72h | QoR-15 at 72 hours after surgery
  the global score of the 15-item Quality of Recovery (QoR-15) questionnaire at 72h after surgery
Number rating score (NRS) | NRS at 24 hours and 72 hours after surgery
  Postoperatvie pain was evaluated using a number rating score (NRS) (0 = no pain, 10 = worst pain possible).
postoperative adverse events | during hospitalization, an average of 2 weeks, assessed up to 30 days
  postoperative adverse events included major adverse cardiovascular events (MACCEs), moderate to severe acute kidney injury (AKI), moderate to severe acute liver injury, reintubation, and postoperative nausea and vomiting (PONV).
chronic pain | at 3 months after surgery
  persistent postoperative pain lasting beyond 3 months

OTHER OUTCOMES:
Postoperative mechanical ventilation | The time from the end of operation to the removal of tracheal intubation, assessed up to 30 days
  The time from the end of operation to the removal of tracheal intubation
hospital length of stay (LOS) | From the date of admission until the date of discharging, assessed up to 30 days
  From the date of admission until the date of discharging
hospital costs | during hospitalization, an average of 2 weeks, assessed up to 30 days
  Total cost of patients during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Data availuable by sending email to corresponding authors